CLINICAL TRIAL: NCT02327273
Title: Randomized, Placebo-Controlled, Double-Blind, Ascending Single and Multiple Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of BMS-963272 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MB006-002
Record Dates: First submitted 2014-12-24; First posted 2014-12-30 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A SAD: BMS-963272 or Placebo (Experimental): BMS-963272 or Placebo oral capsule on specific days
  Interventions: Drug: BMS-963272; Drug: Placebo
- Part B MAD: BMS-963272 or Placebo (Experimental): BMS-963272 or Placebo oral capsule on specific days
  Interventions: Drug: BMS-963272; Drug: Placebo

INTERVENTIONS:
Drug: BMS-963272
Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety profile, tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) following single and multiple oral doses of BMS-963272 in healthy subjects.

DETAILED DESCRIPTION:
Study Classification: Safety, PK/PD

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs and clinical laboratory determinations
* Body Mass Index (BMI) of 27 to 40 kg/m2 inclusive. BMI = weight (kg)/ [height (m)]2
* Females (not of childbearing potential and males, ages 18 to 55 years, inclusive. Female subjects must have documented proof that they are not of childbearing potential
* Azoospermic males and women who are not of child-bearing potential (i.e. are postmenopausal or surgically sterile; see section 3.3.3 for the definition of WOCBP) are exempt from contraceptive requirements. However, women must still undergo pregnancy testing as described in this section

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population
* Any of the following on 12-lead electrocardiogram (ECG) prior to study drug administration, confirmed by repeat.

  i)PR ≥ 210 msec ii)QRS ≥ 120 msec iii)QT ≥ 500 msec iv)QTcF ≥ 450 msec
* Positive urine screen for drugs of abuse
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or HIV-1, -2 antibody
* Moderate anemia (hemoglobin < 11 g/dL for men and < 10 g/dL for women)
* aspartate aminotransferase (AST) > 1.3x ULN
* alanine aminotransferase (ALT) > 1.3x ULN
* Total bilirubin > 1.3x upper limit of normal (ULN)
* estimated glomerular filtration rate (eGFR) < 90 ml/min/1.73 m2 (calculated using CKD-EPI formula)
* HbA1c > 6.5%
* Fasting total cholesterol > 300 mg/dl
* Fasting triglycerides > 400 mg/dl
* Systolic blood pressure > 160 mm Hg and/or diastolic blood pressure > 95 mm Hg, confirmed by repeat measurement
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity).
* History of lactose intolerance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single oral dose of BMS-963272 in healthy overweight and obese subjects is measured by adverse events, Serious adverse events, vital signs, laboratory assessments and ECG | Up to 10 days
Safety and tolerability of multiple oral doses of BMS-963272 in healthy overweight and obese subjects is measured by adverse events, Serious adverse events, vital signs, laboratory assessments and ECG | With in 18 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx